CLINICAL TRIAL: NCT04458519
Title: Randomised Single Blinded Clinical Study of Efficacy of Intranasal Probiotic Treatment to Reduce Severity of Symptoms in COVID19 Infection
Brief Title: Efficacy of Intranasal Probiotic Treatment to Reduce Severity of Symptoms in COVID19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROBCO; 249512 (Other: Health Canada)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2020-07

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; Nasal irrigation; Probiotic; Microbiome; Lactococcus lactis W136
MeSH Terms: conditions — COVID-19 | interventions — Probiotics; Saline Solution

STUDY DESIGN:
Intervention Model Description: Single-blinded, randomized, prospective trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Investigator responsible for product allocation and blinding is not in contact with study participant and will only be made aware of the process of their evolution in case of emergency.
  Study personel in daily contact with the patient are unaware of the patient treatment assignement and are thus blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiorinse (Experimental): Nasal irrigations with Probiorinse (2.4 Billion CFU (Colony-Forming Units) of Lactococcus Lactis W136, (NPN: 80085895)) twice-daily for a period of fourteen days
  Interventions: Other: Probiorinse
- Saline solution (Active Comparator): Nasal irrigations with saline (NeilMed Sinus Rinse, (NPN: 80027142)) twice-daily for a period of fourteen days
  Interventions: Other: Saline solution

INTERVENTIONS:
Other: Probiorinse — Nasal irrigations with probiotic twice-daily for a period of fourteen days
  Other Names: Natural health products; Probiotic
  Arms: Probiorinse
Other: Saline solution — Nasal irrigations with saline-only twice-daily for a period of fourteen days
  Other Names: Natural health product
  Arms: Saline solution

SUMMARY:
Randomised, single-blinded trial. Patients with a diagnosis of COVID-19 infection within the past 96 hours and not requiring hospitalization will be recruited into a trial of BID Nasal irrigation for 14 days, followed by a 14 day observation period. Irrigation will be performed with either Probiorinse probiotic nasal irrigation solution or NeilMed Sinus rinse. Patients will be able to identify their treatments, but study staff will be blinded as to assignment.

DETAILED DESCRIPTION:
BACKGROUND/OBJECTIVE

The potential role of the microbiome in COVID-19 disease remains little explored, yert may offer an unique therapeutic opportunity for its treatment. Airway inflammation and microbiome dysbiosis is present in COVID-19 patients and is related to evolution. The limited information on airway inflammation in COVID-19 suggests greater inflammation, as assessed by serum markers of inflammation, is associated by more severe disease. Late cell-mediated T-cell activation is paradoxically accompanied by TLR expression downregulation, which contributes to dysfunctional immune regulation. Individual predisposition to heightened inflammatory responses may contribute to this.

The investigators believe this early TLR downregulation is an important feature of the disease, allowing the disease to reproduce unchecked and spread during a prolonged asymptomatic shedding period.

Immune-evasion strategies are common to several viral infections such as influenza, respiratory syncytial virus, and human rhinovirus, COVID-19 may exploit this as well.

Lung microbiome data in COVID-19 is limited, but a small dataset of 8 hospitalised cases has been reported from China suggests pulmonary inflammation can be influenced by the microbiome at the time of intubation, arguing the need for a more favorable upper airway microbiome.

Based on the above information, the investigators believe that administration of probiotic bacteria directly to the upper airway via irrigation to patients receiving a diagnosis of COVID-19 will improve the status of the upper airway microbiome and reduce symptom severity and disease in patients with COVID-19 disease not requiring ICU admission or intubation.

The investigators believe intranasally applied 'health-inducing' bacteria will favorably modulate the response to COVID-19 infection, reducing its severity and complications. Probiorinse may exert potentially beneficial effects in COVID-19 infection via two potential and distinct mechanisms:

1. Activation of the innate immune system via enhanced TLR signalling:

   - Abundant TLR ligands present on the probiotic bacterial capsule may counter the downregulation in TLR expression and function seen with COVID-19 infection.
2. Promotion of a 'healthy' microbiome profile in the nasopharynx:

   * Reducing "seeding" the lower respiratory tract with inappropriate bacteria or pathogens.
   * Conditioning inappropriate or excessive immune responses of the airway

The purpose of this clinical trial is thus to compare the safety and validity of intranasal irrigation with Lactococcus lactis W136 with saline nasal irrigation alone in patients with mild COVID-19 infection.

METHODOLOGY

Consent process in the current context of the COVID-19 pandemic: Verbal consent and confirmation of consent in writing or electronically.

Participants will be recruited via posted signs in the COVID-19 clinic and hospital Intranet advertising a research project for individuals diagnosed with COVID-19 infection.

This study will include three (3) periods, which will take the form of telephone calls / email contacts:

1. Eligibility determination period (Day 0)
2. Treatment period (Day 1 to Day 14): Probiorinse or Saline solution
3. Follow-up period (Day 21 and Day 28)

STATISTICAL ANALYSIS

Analysis population:

The primary analysis population for the efficacy endpoints will be the randomized ITT population which includes all patients who have been allocated to a randomized treatment regardless of whether the treatment kit was used or not. The efficacy analyses will be conducted according to the treatment to which they were randomized.

The analysis population for safety endpoints is defined as all patients exposed to study medication, regardless of the amount of treatment administered. The safety analyses will be conducted according to the treatment patients actually received. The treatment emergent period is defined as the time from the first administration of study medication to Day 14 of post treatment period.

Data Analysis:

The following null hypothesis and alternative will be tested for the Probiorinse arm against NeilMed Sinus Rinse:

* H0: No treatment difference between Probiorinse and NeilMed Sinus Rinse.
* H1: There is a treatment difference between Probiorinse and NeilMed Sinus Rinse

Descriptive statistics including number of subjects mean, standard error, and least squares (LS) means will be provided. In addition, difference in LS means and the corresponding 95% confidence intervals (CI) will be provided along with the p-values.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-59 years
* Positive diagnosis of COVID-19 infection less than 96 hours
* Characteristic respiratory symptoms present but no more than mild to moderate
* No need for oxygen
* Temperature less than 38.0 ºC
* Not presently being considered for hospitalisation or ICU admission
* Able to perform nasal irrigation
* Able to provide consent
* Able to communicate with the study team by phone, text or email

Exclusion Criteria:

* Patients with pre-existing conditions or demographic features placing them at increased risk of complications from COVID10 infection will not be included in this study. These will be considered exclusion factors, thus individuals will be questioned as to the presence or these factors during their telephone screening.
* Respiratory disorders:

  * Asthma, Pre-existing COPD, bronchiectasis or cystic fibrosis
* Hypertension
* Cardiovascular disease:

  * Rhythm disturbances, recent (less than 6 months), angina pectoris cardiac insufficiency
* Diabetes
* Immunosuppressed patients (other than COVID-19 induced)

  * Primary immune deficiencies such as hypogammaglobulinemia or common variable immune deficiency (CVID)
  * Chemotherapy depressing the immune system
  * Immune suppressing medications such as prednisone, Imuran, or TNF inhibitors, or anti-rejection transplant drugs.
  * Solid organ transplant
* Cancer under treatment or within five years (except basocellular skin cancers)
* Pregnant or breastfeeding women or women unwilling to practice contraception as outlined in the study protocol for the duration of the study period.
* Allergy to milk or its derivatives

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Change in severity of COVID-19 infection | 4 weeks
  Change in severity of COVID-19 infection as assessed by number of days with any symptoms of COVID-19 infection greater than or equal to 35 as measured on VAS scale as assessed at the 28 day endpoint.

SECONDARY OUTCOMES:
Number of days with any symptom of anosmia | 4 weeks
  Number of days with any symptom of anosmia
Maximal intensity attained in overall assessment of symptoms of COVID-19 infection as measured on Visual Analogue Scale (VAS). | 4 weeks
  Maximal intensity attained in overall assessment of symptoms of COVID-19 infection as measured on Visual Analogue Scale (VAS). VAS scale from 0 to 100, with a higher score indicating a worse outcome.
Number of days where rescue medication is required | 4 weeks
  Number of days where rescue medication is required

CONTACTS AND LOCATIONS:
Overall Officials: Martin Y Desrosiers, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu J, Li S, Liu J, Liang B, Wang X, Wang H, Li W, Tong Q, Yi J, Zhao L, Xiong L, Guo C, Tian J, Luo J, Yao J, Pang R, Shen H, Peng C, Liu T, Zhang Q, Wu J, Xu L, Lu S, Wang B, Weng Z, Han C, Zhu H, Zhou R, Zhou H, Chen X, Ye P, Zhu B, Wang L, Zhou W, He S, He Y, Jie S, Wei P, Zhang J, Lu Y, Wang W, Zhang L, Li L, Zhou F, Wang J, Dittmer U, Lu M, Hu Y, Yang D, Zheng X. Longitudinal characteristics of lymphocyte responses and cytokine profiles in the peripheral blood of SARS-CoV-2 infected patients. EBioMedicine. 2020 May;55:102763. doi: 10.1016/j.ebiom.2020.102763. Epub 2020 Apr 18. PMID 32361250
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Liu Y, Yan LM, Wan L, Xiang TX, Le A, Liu JM, Peiris M, Poon LLM, Zhang W. Viral dynamics in mild and severe cases of COVID-19. Lancet Infect Dis. 2020 Jun;20(6):656-657. doi: 10.1016/S1473-3099(20)30232-2. Epub 2020 Mar 19. No abstract available. PMID 32199493
- [Background] Shen Z, Xiao Y, Kang L, Ma W, Shi L, Zhang L, Zhou Z, Yang J, Zhong J, Yang D, Guo L, Zhang G, Li H, Xu Y, Chen M, Gao Z, Wang J, Ren L, Li M. Genomic Diversity of Severe Acute Respiratory Syndrome-Coronavirus 2 in Patients With Coronavirus Disease 2019. Clin Infect Dis. 2020 Jul 28;71(15):713-720. doi: 10.1093/cid/ciaa203. PMID 32129843
- See also: Study publication (Pre-print) — https://www.medrxiv.org/content/10.1101/2021.04.18.21255699v1.full